CLINICAL TRIAL: NCT03509636
Title: An Open-Label Study to Assess the Efficacy And Safety of Poly(ADP-ribose) Polymerase Inhibitor Fluzoparib（SHR3162）in Patients With Relapsed High-grade Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer and BRCA1/2 Mutation
Brief Title: A Study of Fluzoparib（SHR-3162）in BRCA1/2-mutant Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-FZPL-Ⅰb-OC
Record Dates: First submitted 2018-02-25; First posted 2018-04-26 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Fluzoparib capsule
  Interventions: Drug: Fluzoparib

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib capsule will be given twice daily orally
  Other Names: SHR-3162

SUMMARY:
This is a multicenter， open-label study to evluate the efficacy and safety of a novel PARP 1/2 inhibitor fluzoparib （SHR-3162）in BRCA1/2-mutant Relapsed Ovarian Cancer.

DETAILED DESCRIPTION:
Fluzoparib (SHR-3162) is an orally available, small molecule inhibitor of poly-adenosine diphosphate [ADP] ribose polymerase (PARP) 1/2 being developed for treatment of BRCA1/2-mutant solid tumor. The tolerability, safety and PK of fluzoparib has been evaluated in Phase 1 study. An oral formulation is the focus of current development efforts.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of high grade serous or Grade 2/3 endometrioid epithelial ovarian, fallopian tube, or primary peritoneal cancer；
* Confirmed documented BRCA1/2 mutation;
* Received 2~4 prior chemotherapy regimens. Non-chemotherapy regimens and maintenance therapies administered as single agent treatment will not count as a chemotherapy regimen；
* Relapsed/progressive disease as confirmed by radiologic assessment；
* Have measurable disease as defined by RECIST v1.1.

Exclusion Criteria:

* Any previous treatment with a PARP inhibitor;
* Patient with any other malignancy which has been active or treated within the previous 5 years;
* Patients with symptomatic uncontrolled brain metastases;
* Patients unable to swallow orally administered medication.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
ORR by RECIST v1.1 | every 8 weeks (±7 days) of treatment
  Objective response rate

SECONDARY OUTCOMES:
DoR | study data collection expected to last for ~2 years
  Duration of response
PFS | expected to last for ~2 years
  Progression free survival
Response rate by GCIG CA-125 | every 8 weeks (±7 days) of treatment expected to last for ~2 years
  Response rate per GCIG CA-125
OS | study data collection expected to last for ~2 years
  Overall suvival
Incidence of adverse events, clinical laboratory abnormalities, and dose modifications | Every day starting with signing of consent until 30 days after discontinuation of treatment
  per CTC AE 4.03
Trough (Cmin) level of fluzoparib concentrations | Cycle 1 to cycle 4(each cycle is 28 days)
  Cssmin of fluzoparib concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided